CLINICAL TRIAL: NCT07367230
Title: Effects of Elastic Band-Resisted Plyometric Training on Jump Performance in Young Male Soccer Players: A Randomized Controlled Trial
Brief Title: Elastic Band-Resisted Plyometric Training in Young Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serkan özgür (Other)
Responsible Party: Sponsor-Investigator, Serkan özgür, Lecturer, Manisa Celal Bayar University
Organization: Manisa Celal Bayar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20.478.486-3318,30/07/2025
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Athletic Performance; Plyometric Exercises; Physical Conditioning, Human
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three parallel groups: elastic band-resisted plyometric training (EBPT, n=10), traditional plyometric training (PLT, n=11), or control (CON, n=12). All participants remained in their assigned groups throughout the 6-week intervention period. Both intervention groups received plyometric training twice weekly, while the control group continued regular soccer training only.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elastic Band-Resisted Plyometric Training (EBPT) (Experimental): Participants performed plyometric exercises with elastic band resistance for 6 weeks, 2 sessions per week
  Interventions: Behavioral: Elastic Band-Resisted Plyometric Training
- Traditional Plyometric Training (PLT) (Active Comparator): Participants performed traditional plyometric exercises without elastic band resistance for 6 weeks, 2 sessions per week,
  Interventions: Behavioral: Traditional Plyometric Training
- Control (CON) (Active Comparator): Participants continued their regular soccer training without any additional plyometric exercises during the 6-week intervention period.
  Interventions: Other: Regular Soccer Training (No Intervention)

INTERVENTIONS:
Behavioral: Elastic Band-Resisted Plyometric Training — Participants performed plyometric exercises (squat jumps, countermovement jumps, drop jumps, and single-leg jumps) with elastic band resistance providing additional load during the concentric phase. Training was conducted twice weekly for 6 weeks, with 124-224 foot contacts per session.
  Arms: Elastic Band-Resisted Plyometric Training (EBPT)
Behavioral: Traditional Plyometric Training — Participants performed the same plyometric exercises (squat jumps, countermovement jumps, drop jumps, and single-leg jumps) without elastic band resistance. Training was conducted twice weekly for 6 weeks, with 124-224 foot contacts per session.
  Arms: Traditional Plyometric Training (PLT)
Other: Regular Soccer Training (No Intervention) — Participants continued their routine soccer training program without any additional plyometric exercises during the 6-week study period.
  Arms: Control (CON)

SUMMARY:
This randomized controlled trial investigated the effects of elastic band-resisted plyometric training (EBPT) on jump performance in young male soccer players. Thirty-three youth soccer players aged 14-15 years were randomly assigned to one of three groups: elastic band-resisted plyometric training (EBPT, n=10), traditional plyometric training (PLT, n=11), or control (CON, n=12). Both training groups completed a 6-week intervention consisting of 2 sessions per week with 350-800 foot contacts per session. The primary outcome was countermovement jump without arm swing (CMJ-NS) height. Secondary outcomes included squat jump (SJ), countermovement jump with arm swing (CMJ-AS), single-leg vertical jumps for dominant (SVJ-D) and non-dominant (SVJ-ND) legs, take-off velocity, and peak power. Assessments were conducted at baseline and post-intervention. The study aimed to determine whether adding elastic band resistance to plyometric exercises provides superior training adaptations compared to traditional plyometric training for enhancing lower-limb explosive power in young athletes.

ELIGIBILITY:
Inclusion Criteria:

* Male soccer players aged 14-15 years
* Member of a registered soccer academy
* Minimum 2 years of soccer training experience
* Regular participation in team training (at least 3 sessions per week)
* No participation in systematic plyometric training in the previous 6 months
* Written informed consent from parent/guardian

Exclusion Criteria:

* Current musculoskeletal injury or pain
* History of lower extremity surgery in the past 12 months
* Any cardiovascular or respiratory condition that contraindicates high-intensity exercise
* Participation in other training intervention studies
* Inability to attend at least 80% of training sessions

Ages: 14 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Countermovement Jump Without Arm Swing (CMJ-NS) Height | Baseline and 6 weeks (post-intervention)
  Vertical jump height measured during countermovement jump without arm swing, assessed using a portable force platform.

SECONDARY OUTCOMES:
Squat Jump (SJ) Height | Baseline and 6 weeks
  Vertical jump height measured during squat jump using a portable force platform.
Countermovement Jump With Arm Swing (CMJ-AS) Height | Baseline and 6 weeks
  Vertical jump height measured during countermovement jump with arm swing using a portable force platform.
Single-Leg Vertical Jump - Dominant Leg (SVJ-D) Height | Baseline and 6 weeks
  Vertical jump height measured during single-leg jump from the dominant leg using a portable force platform.
Single-Leg Vertical Jump - Non-Dominant Leg (SVJ-ND) Height | Baseline and 6 weeks
  Vertical jump height measured during single-leg jump from the non-dominant leg using a portable force platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Guzeltepe sport club facility, Izmir, Guzeltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No